CLINICAL TRIAL: NCT04303195
Title: A Phase 2 Randomized, Double-blind, Placebo-Controlled, Parallel-Group Study, of the Safety and Efficacy of NG101 Administered Orally to Patients With Gastroparesis
Brief Title: A Study to Evaluate the Safety and Efficacy of NG101 in Adult Participants With Symptomatic Diabetic or Idiopathic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurogastrx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NG101-201
Record Dates: First submitted 2020-02-12; First posted 2020-03-10 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Gastroparesis; Idiopathic Gastroparesis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NG101 - 5 mg (Experimental): NG101 5 mg, capsules, orally, QID (4 times a day) for up to 12 weeks
  Interventions: Drug: NG101
- NG101 - 10 mg (Experimental): NG101 10 mg, capsules, orally, QID (4 times a day) for up to 12 weeks
  Interventions: Drug: NG101
- NG101 - 20 mg (Experimental): NG101 20 mg, capsules, orally, QID (4 times a day) for up to 12 weeks
  Interventions: Drug: NG101
- Placebo (Placebo Comparator): Placebo-matching, capsules, orally, QID (4 times a day) for up to 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NG101 — Capsules
  Other Names: metopimazine mesylate
  Arms: NG101 - 10 mg; NG101 - 20 mg; NG101 - 5 mg
Drug: Placebo — Capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of various dose levels of NG101 compared with placebo in adult participants with gastroparesis during 12 weeks of treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group , placebo-controlled, multicenter US-based study to evaluate the safety and efficacy of 3 dose levels of NG101 (Metopimazine mesylate) compared with placebo in participants with diabetic or idiopathic gastroparesis.

The study will enroll approximately 140 participants. Following the Screening Period, there is a 2-week Pretreatment Period during which participants will complete an electronic daily diary. Participants eligible for the clinical study will be randomly assigned (in a 1:1:1:1 ratio) to receive either NG101 5 mg, 10 mg, or 20 mg, or matching placebo during a 12-week Treatment Period. All participants will be asked to take one capsule 30 minutes before a meal 3 times a day and 30 minutes before bedtime for a total of 4 capsules daily (QID). The total duration of the study for each participant will be approximately 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with diabetic or idiopathic gastroparesis
* Symptoms consistent with gastroparesis (nausea, vomiting, early satiety, post-prandial fullness, and abdominal pain)
* Documented evidence of no mechanical obstruction
* Delayed gastric emptying as demonstrated by gastric scintigraphy or breath test

Exclusion Criteria:

* Uncontrolled diabetes (defined as HgbA1c > 10%)
* Severe postural symptoms or evidence of unexplained recurrent dizziness
* Participant has received and tolerated domperidone and showed no notable symptomatic improvement in gastroparesis symptoms
* Participant has had endoscopic pyloric injections of botulinum toxin within the 6 months prior to the Screening Visit.
* Participant engages in daily recreational use of marijuana
* Prolactin levels > 2 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (82):
- United States (82):
  - Digestive Health Specialists, Dothan, Alabama
  - G & L Research, LLC, Foley, Alabama
  - East View Medical Research, Mobile, Alabama
  - Phoenix Medical Group, Peoria, Arizona
  - Phoenix Clinical LLC, Phoenix, Arizona
  - Del Sol Research Management, Tucson, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - GW Research, Inc, Chula Vista, California
  - Precision Research Institute, LLC, Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Diagnamics Inc., Encinitas, California
  - Paragon Rx Clinical, Inc, Garden Grove, California
  - United Clinical Research, Irvine, California
  - Prime Care Clinical Rsearch, Laguna Hills, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - Angel City Research, Los Angeles, California
  - United Clinical Research, Murrieta, California
  - Diabetes Medical Center of California, Northridge, California
  - Precision Research Institute, San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Innovative Research of West Florida, Clearwater, Florida
  - Innovation Medical Group, LLC., Fort Lauderdale, Florida
  - ENCORE Borland-Grover Clinical Research, Jacksonville, Florida
  - ClinCloud, LLC, Maitland, Florida
  - Verus Clinical Research, Corp, Miami, Florida
  - APF Research, LLC, Miami, Florida
  - Panax Clinical Research, Miami, Florida
  - International Research Associates LLC, Miami, Florida
  - PharmaSouth Research, Miami, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - AES - DRS - Synexus Clinical Research US, Inc. - St. Petersburg, Pinellas Park, Florida
  - Avita Clinical Research, Tampa, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - IResearch Atlanta LLC, Decatur, Georgia
  - Claude Mandel Medical Center, Chicago, Illinois
  - Medisphere Medical Research Center LLC, Evansville, Indiana
  - Indiana University Hospital, Indianapolis, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - West Glen GI, Shawnee Mission, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - Clinical Trials of America, West Monroe, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - KLEO Health & Research, Missoula, Montana
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Digestive Disease Specialists, Las Vegas, Nevada
  - Lovelace Respiratory Rsearch Institute, Albuquerque, New Mexico
  - Synexus Clinical Research, New York, New York
  - Tandem Clinical Research GI, LLC, New York, New York
  - Javara Research, Charlotte, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - Carolina Digestive Diseases, Greenville, North Carolina
  - Dayton Gastroenterology Inc., Beavercreek, Ohio
  - Hometown Urgent Care and Research, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Draelos Metabolic Center, Edmond, Oklahoma
  - Options Health Research, Tulsa, Oklahoma
  - Transsouth Healthcare PC, Jackson, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Avant Research Associates, Austin, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Sante Clinical Research, Kerville, Texas
  - Rio Grande Gastroenterology, McAllen, Texas
  - DM Clinical Research Solutions PC, Pearland, Texas
  - AES - DRS - Synexus Clinical Research US, Inc. - Plano, Plano, Texas
  - Sun Research, San Antonio, Texas
  - Southern Star Research Institute, San Antonio, Texas
  - Synexus Clinical Research, San Antonio, Texas
  - Horizon Clinical Research- Tomball, Tomball, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Velocity Clinical Research Spokane, Spokane, Washington

REFERENCES:
- [Derived] Loesch J, Hamza E, Pasricha PJ, Nee J, Cline M, MacDougall J, Simons M, Brown JT, Garg S, Hoscheit M, Gabbard S, De Colle C, Lembo A. A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Metopimazine Mesylate (NG101) in Participants With Gastroparesis. Am J Gastroenterol. 2026 Feb 1;121(2):534-544. doi: 10.14309/ajg.0000000000003534. Epub 2025 May 14. PMID 40367443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with symptomatic idiopathic or diabetic gastroparesis took part in the study at 51 investigative sites in the United States from 01 August 2020 to 25 February 2023
Pre-assignment Details: Participants eligible for the study were randomized in a 1:1:1:1 ratio to receive either NG101 treatment arms of 5 mg, 10 mg, or 20 mg, or matching placebo during a 12-week Treatment Period. Randomization was stratified on the following factors: gastroparesis etiology (diabetes vs idiopathic), sex (male vs female), and current cannabinoid use (yes vs no).
Period: Overall Study
Arm/Group | NG101 - 5 mg | NG101 - 10 mg | NG101 - 20 mg | Placebo
Started | 40 | 41 | 40 | 40
Completed | 35 | 35 | 31 | 33
Not Completed | 5 | 6 | 9 | 7
Not completed — Adverse Event | 1 | 3 | 7 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 4
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 1
Not completed — No study drug administered or protocol deviation | 0 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: This study included a Screening Period of up to 6 weeks and a 2-week Pretreatment Period. Following successful completion of the Pretreatment Period, participants eligible for the clinical study were randomized in a 1:1:1:1 ratio to receive either NG101 5 mg, 10 mg, or 20 mg, or matching placebo during a 12-week Treatment Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | NG101 - 5 mg | NG101 - 10 mg | NG101 - 20 mg | Placebo | Total
Number analyzed (Participants) | 40 | 41 | 40 | 40 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 30 | 29 | 123
  >=65 years | 8 | 9 | 10 | 11 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (11.5) | 53.7 (11.26) | 55.7 (13.50) | 55.4 (14.19) | 54.5 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 33 | 33 | 133
  Male | 7 | 7 | 7 | 7 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 20 | 20 | 16 | 73
  Not Hispanic or Latino | 23 | 21 | 20 | 24 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 9 | 4 | 9 | 23
  White | 39 | 32 | 33 | 30 | 134
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 40 | 40 | 161
Gastroparesis etiology [Count of Participants; unit: Participants]
  Diabetic | 18 | 19 | 19 | 17 | 73
  Idiopathic | 22 | 22 | 21 | 23 | 88
Cannabinoid use [Count of Participants; unit: Participants]
  Yes | 4 | 3 | 3 | 5 | 15
  No | 36 | 38 | 37 | 35 | 146

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Nausea Severity Score
Description: Change from Baseline at Weeks 7 through 12 (average) as measured by the Diabetic and Idiopathic Gastroparesis Symptoms Daily Diary (DIGS-DD). Participants were asked to rate their symptoms at their worst in the past 24 hours using a 0 to 10-point numeric rating scale (NRS). A score of 0 indicates no symptoms and a score of 10 indicates the worst possible symptoms. For each week in the 2-week Pretreatment Period, the 12-week Treatment Period, and the 2-week Follow-up Period, a participant's score for that week was the mean of the daily scores for that week. A negative change from baseline indicates improvement.
Time Frame: Baseline to Week 12
Population: Per Protocol population included all participants in the Intent-To-Treat Population (all enrolled participants who were randomized) who do not have any major protocol deviations that would affect efficacy as determined by the study team.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NG101 - 5 mg | NG101 - 10 mg | NG101 - 20 mg | Placebo
Number analyzed (Participants) | 37 | 33 | 33 | 33
units on a scale | -3.55 (0.331) | -3.65 (0.0348) | -3.43 (0.348) | -2.83 (0.347)
Statistical Analysis 1: Comparison: NG101 - 5 mg vs Placebo; Test type: Superiority; p = 0.1350, ANOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.67 to 0.23], Standard Error of Mean 0.479
Statistical Analysis 2: Comparison: NG101 - 10 mg vs Placebo; Test type: Superiority; p = 0.0997, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.79 to 0.16], Standard Error of Mean 0.493
Statistical Analysis 3: Comparison: NG101 - 20 mg vs Placebo; Test type: Superiority; p = 0.2195, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-1.58 to 0.37], Standard Error of Mean 0.492

2. Secondary Outcome: Change From Baseline in Early Satiety Severity Score
Description: Change from baseline at Weeks 7 through 12 (average) as measured by the Diabetic and Idiopathic Gastroparesis Symptoms Daily Diary (DIGS-DD) for early satiety severity score.
  Participants were asked to rate their symptoms at their worst in the past 24 hours using a 0 to 10-point numeric rating scale (NRS). A score of 0 indicates no symptoms and a score of 10 indicates the worst possible symptoms. For each week in the 2-week Pretreatment Period, the 12-week Treatment Period, and the 2-week Follow-up Period, a participant's score for that week was the mean of the daily scores for that week. A negative change from baseline indicates improvement.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NG101 - 5 mg | NG101 - 10 mg | NG101 - 20 mg | Placebo
Number analyzed (Participants) | 37 | 33 | 33 | 33
units on a scale | -3.02 (0.343) | -3.23 (0.360) | -2.64 (0.362) | -2.89 (0.361)
Statistical Analysis 1: Comparison: NG101 - 5 mg vs Placebo; Test type: Superiority; p = 0.7944, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-1.11 to 0.85], Standard Error of Mean 0.498
Statistical Analysis 2: Comparison: NG101 - 10 mg vs Placebo; Test type: Superiority; p = 0.4956, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.36 to 0.66], Standard Error of Mean 0.510
Statistical Analysis 3: Comparison: NG101 - 20 mg vs Placebo; Test type: Superiority; p = 0.6260, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.76 to 1.26], Standard Error of Mean 0.511

3. Secondary Outcome: Change From Baseline in Postprandial Fullness Severity Score
Description: Change from baseline at Weeks 7 through 12 (average) as measured by patient's daily diary entries during participation in the study for postprandial fullness severity score.
  Participants were asked to rate their symptoms at their worst in the past 24 hours using a 0 to 10-point numeric rating scale (NRS). A score of 0 indicates no symptoms and a score of 10 indicates the worst possible symptoms. For each week in the 2-week Pretreatment Period, the 12-week Treatment Period, and the 2-week Follow-up Period. A negative change from baseline indicates improvement.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NG101 - 5 mg | NG101 - 10 mg | NG101 - 20 mg | Placebo
Number analyzed (Participants) | 37 | 33 | 33 | 33
units on a scale | -2.94 (0.373) | -2.96 (0.392) | -2.67 (0.393) | -2.87 (0.394)
Statistical Analysis 1: Comparison: NG101 - 5 mg vs Placebo; Test type: Superiority; p = 0.8866, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-1.15 to 1.00], Standard Error of Mean 0.543
Statistical Analysis 2: Comparison: NG101 - 10 mg vs Placebo; Test type: Superiority; p = 0.8699, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-1.19 to 1.01], Standard Error of Mean 0.558
Statistical Analysis 3: Comparison: NG101 - 20 mg vs Placebo; Test type: Superiority; p = 0.7297, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.91 to 1.29], Standard Error of Mean 0.556

4. Secondary Outcome: Change From Baseline in Abdominal Pain Severity Score
Description: as for outcome 3
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NG101 - 5 mg | NG101 - 10 mg | NG101 - 20 mg | Placebo
Number analyzed (Participants) | 37 | 33 | 33 | 33
units on a scale | -2.65 (0.280) | -2.69 (0.292) | -2.19 (0.293) | -2.70 (0.295)
Statistical Analysis 1: Comparison: NG101 - 5 mg vs Placebo; Test type: Superiority; p = 0.9034, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.76 to 0.86], Standard Error of Mean 0.409
Statistical Analysis 2: Comparison: NG101 - 10 mg vs Placebo; Test type: Superiority; p = 0.9742, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.68 to 0.63], Standard Error of Mean 0.330
Statistical Analysis 3: Comparison: NG101 - 20 mg vs Placebo; Test type: Superiority; p = 0.2235, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.31 to 1.33], Standard Error of Mean 0.417

5. Secondary Outcome: Change From Baseline in Discrete Episodes of Vomiting
Description: Change from baseline at Weeks 7 through 12 (average) as measured by patient's daily diary entries during participation in the study for the number of discrete episodes of vomiting.
  Participants were asked to record the number of episodes of vomiting in the past 24 hours. Each episode counts as "1". A negative change from baseline indicates improvement.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NG101 - 5 mg | NG101 - 10 mg | NG101 - 20 mg | Placebo
Number analyzed (Participants) | 37 | 33 | 33 | 33
units on a scale | -0.42 (0.081) | -0.50 (0.085) | -0.40 (0.085) | -0.31 (0.085)
Statistical Analysis 1: Comparison: NG101 - 5 mg vs Placebo; Test type: Superiority; p = 0.3567, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.34 to 0.12], Standard Error of Mean 0.118
Statistical Analysis 2: Comparison: NG101 - 10 mg vs Placebo; Test type: Superiority; p = 0.1129, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.43 to 0.05], Standard Error of Mean 0.120
Statistical Analysis 3: Comparison: NG101 - 20 mg vs Placebo; Test type: Superiority; p = 0.4590, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.33 to 0.15], Standard Error of Mean 0.120

6. Secondary Outcome: Change From Baseline in 3-symptom Severity Score
Description: Change from baseline at Weeks 7 through 12 (average) as measured by patient's daily diary entries during participation in the study for 3-symptom severity score.
  Participants were asked to rate their symptoms at their worst in the past 24 hours using a 0 to 10-point numeric rating scale (NRS). A score of 0 indicates no symptoms and a score of 10 indicates the worst possible symptoms. For each week, the 3-symptom severity score is the average of the mean daily scores of nausea, early satiety, and postprandial fullness severity scores. A negative change from baseline indicates improvement.
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NG101 - 5 mg | NG101 - 10 mg | NG101 - 20 mg | Placebo
Number analyzed (Participants) | 37 | 33 | 33 | 33
units on a scale | -3.16 (0.334) | -3.28 (0.351) | -2.92 (0.352) | -2.85 (0.352)
Statistical Analysis 1: Comparison: NG101 - 5 mg vs Placebo; Test type: Superiority; p = 0.5250, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-1.27 to 0.65], Standard Error of Mean 0.485
Statistical Analysis 2: Comparison: NG101 - 10 mg vs Placebo; Test type: Superiority; p = 0.3991, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.41 to 0.56], Standard Error of Mean 0.498
Statistical Analysis 3: Comparison: NG101 - 20 mg vs Placebo; Test type: Superiority; p = 0.9006, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-1.05 to 0.92], Standard Error of Mean 0.497

7. Secondary Outcome: Change From Baseline in 4-symptom Severity Score
Description: Change from baseline at Weeks 7 through 12 (average) as measured by patient's daily diary entries during participation in the study for 4-symptom severity score.
  Participants were asked to rate their symptoms at their worst in the past 24 hours using a 0 to 10-point numeric rating scale (NRS). A score of 0 indicates no symptoms and a score of 10 indicates the worst possible symptoms. For each week, the 4-symptom severity score is the average of the mean daily scores of nausea, early satiety, postprandial fullness, and abdominal pain severity scores. A negative change from baseline indicates improvement
Time Frame: Baseline to Week 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NG101 - 5 mg | NG101 - 10 mg | NG101 - 20 mg | Placebo
Number analyzed (Participants) | 37 | 33 | 33 | 33
units on a scale | -3.04 (0.306) | -3.14 (0.321) | -2.74 (0.322) | -2.81 (0.321)
Statistical Analysis 1: Comparison: NG101 - 5 mg vs Placebo; Test type: Superiority; p = 0.6009, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-1.11 to 0.64], Standard Error of Mean 0.444
Statistical Analysis 2: Comparison: NG101 - 10 mg vs Placebo; Test type: Superiority; p = 0.4654, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-1.23 to 0.56], Standard Error of Mean 0.454
Statistical Analysis 3: Comparison: NG101 - 20 mg vs Placebo; Test type: Superiority; p = 0.8842, ANCOVA — The threshold for statistical significance was p = 0.05; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.83 to 0.97], Standard Error of Mean 0.455

ADVERSE EVENTS:
Time Frame: From study start (randomization) through the End of Study/Safety Visit (approximately 14 weeks)
Description: All AEs ad SAEs were collected starting from signature of ICF until the End of Study/Safety Follow-up Visit.
  Note that in the placebo arm, 40 participants were randomized and included in the intent-to-treat efficacy analyses, but only 39 participants received at least one dose of placebo. Data is provided for all 40 randomized participants.
Arm/Group | NG101 - 5 mg | NG101 - 10 mg | NG101 - 20 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/41 | 1/40 | 0/40
Other Adverse Events (participants affected / at risk) | 15/40 | 12/41 | 21/40 | 14/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NG101 - 5 mg (N=40) | NG101 - 10 mg (N=41) | NG101 - 20 mg (N=40) | Placebo (N=40)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NG101 - 5 mg (N=40) | NG101 - 10 mg (N=41) | NG101 - 20 mg (N=40) | Placebo (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 1 | 2 | 0
Tachycrdia (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 1 | 1 | 1
Coronavirus infection (Infections and infestations) | 1 | 2 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Pustle (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 3 | 3 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Galactorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT04303195/Prot_SAP_000.pdf